CLINICAL TRIAL: NCT06550986
Title: False Lumen Treatment for Prevention of Aortic Growth Using Shape Memory Polymer - First-in-Human Study
Acronym: FLAGSHIP_NZL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shape Memory Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD1043
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: Intervention (Experimental): Device: False Lumen Embolization System Device: IMPEDE-FX RapidFill
  Interventions: Device: False Lumen Embolization System, IMPEDE-FX RapidFill

INTERVENTIONS:
Device: False Lumen Embolization System, IMPEDE-FX RapidFill — Embolization of the false lumen of an aortic dissection

SUMMARY:
To determine the safety and feasibility of the investigational product to reduce aortic dissection false lumen perfusion.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* A candidate for false lumen (FL) embolization with a type B dissection, and no prior primary entry tear/TL treatment, OR
* A candidate for FL embolization with a type B or type A dissection, in whom the primary entry tear/TL was treated in a previous procedure, and is now presenting with a FL requiring treatment.

Exclusion Criteria:

* An inability to provide informed consent.
* Enrolled in another clinical study other than a registry.
* Hyperacute or acute aortic dissection (<15 days from symptom onset).
* Untreated or uncovered primary entry/reentry tear proximal to left subclavian artery (before FL treatment with the investigational product).
* Vascular disease, aortic rupture, and/or anatomy and/or dissection membrane condition that precludes the safe access and positioning of an introducer sheath and delivery (and expansion) of the investigational product into the FL.
* Prior treatment of the FL.
* Planned use of investigational devices to treat the primary entry tear and/or TL.
* Absence of/inability to create a reentry tear/fenestration adequately positioned and large enough to allow introducer sheath access into the FL.
* Planned use of FL embolic devices other than the investigational product.
* Prior abdominal aortic aneurysm (AAA) treatment.
* Planned concomitant major surgery (e.g., gastrointestinal surgery).
* Diagnosed or suspected congenital degenerative connective tissue disease (e.g., Marfan's or Ehler-Danlos syndrome).
* Coagulopathy or uncontrolled bleeding disorder.
* Serum creatinine level >220 µmol/L (within 90 days prior to the procedure).
* Cerebrovascular accident within 90 days prior to the procedure.
* Myocardial infarction and/or major heart surgery within 90 days prior to the procedure.
* Atrial fibrillation that is not well rate controlled.
* Unable or unwilling to comply with study follow-up requirements.
* Life expectancy of <2 years postprocedure.
* Known hypersensitivity or contraindication to platinum, iridium, or polyurethane.
* A condition that inhibits radiographic visualization during the study procedure and planned follow-up imaging.
* History of allergy to contrast medium that cannot be managed medically.
* Uncontrolled comorbid medical condition, including mental health issues, that, in the opinion of the investigator, would adversely affect participation in the study.
* Participant is planning to become pregnant or is currently pregnant or lactating. For participants of child-bearing potential, based on a positive pregnancy test within 7 days prior to the procedure or refusal to use a medically accepted method of birth control for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Technical success | Immediately after the intervention
  Delivery and implantation of the investigational product implant to the false lumen
Major adverse events | 30 days
  Incidence of device/procedure-related major adverse events

SECONDARY OUTCOMES:
All-cause mortality and dissection-related mortality | 2 years
  Incidence of all-cause mortality and dissection-related mortality
Serious adverse events | 2 years
  Incidence of device/procedure-related serious adverse events
Change in false lumen thrombosis from baseline | 2 years
  Change in false lumen thrombosis from baseline
Change in true lumen/aorta size ratio from baseline | 2 years
  Change in true lumen/aorta size ratio from baseline
Change in aorta size from baseline | 2 years
  Change in aorta size from baseline
Rate of dissection-related reinterventions | 2 years
  Rate of dissection-related reinterventions

CONTACTS AND LOCATIONS:
Locations (1):
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No